CLINICAL TRIAL: NCT01465802
Title: ARCHER 1042: A PHASE 2 STUDY OF DACOMITINIB IN ADVANCED NON-SMALL CELL LUNG CANCER (POST-CHEMOTHERAPY OR SELECT FIRST LINE PATIENTS) TO EVALUATE PROPHYLACTIC INTERVENTION ON DERMATOLOGIC AND GASTROINTESTINAL ADVERSE EVENTS AND PATIENT REPORTED OUTCOMES
Brief Title: Study Of Dacomitinib (PF-00299804) In Advanced NSCLC Patients (Post Chemo Or Select First Line) To Evaluate Prophylactic Intervention On Derm And GI AEs And PRO
Acronym: ARCHER 1042
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A7471042
Record Dates: First submitted 2011-10-20; First posted 2011-11-07 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: non-small cell lung cancer; advanced; previously treated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib; Doxycycline; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort I (Experimental): Arm A: Dacomitinib 45 mg orally daily on a continuous schedule until disease progression, toxicity, death or withdrawal of consent Doxycycline placebo orally BID for 4 weeks Arm B: Dacomitinib 45 mg orally daily on a continuous schedule until disease progression, toxicity, death or withdrawal of consent Doxycycline 100 mg orally BID for 4 weeks
  Interventions: Drug: Dacomitinib; Drug: Doxycycline
- Cohort II (Experimental): Dacomitinib 45 mg orally daily on a continuous schedule until disease progression, toxicity, death or withdrawal of consent Topical alclometasone diproprionate cream 0.05% applied to face, hands, feet, neck, back and chest at bedtime for 4 weeks VSL#3 probiotic 4 capsules orally daily or 1 sachet orally daily for up to 5 weeks (starting between Day minus 7 to Day minus 4 and continuing through Day 28)
  Interventions: Drug: Dacomitinib; Drug: Probiotic; Drug: Alclometasone cream
- Cohort III (Experimental): Cohort III is an interrupted dosing schedule of dacomitinib in the first cycle only
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Dacomitinib 45 mg orally daily on a continuous schedule until disease progression, toxicity, death or withdrawal of consent
  Arms: Cohort I; Cohort II
Drug: Dacomitinib — Dacomitinib 45 mg orally daily on a continuous schedule for the first 10 days in Cycle 1, followed by 4 days off treatment, followed by continuous daily dosing until disease progression, toxicity, death or withdrawal of consent
  Arms: Cohort III
Drug: Doxycycline — Doxycycline or Doxycycline placebo BID for 4 weeks
  Arms: Cohort I
Drug: Probiotic — VSL#3 probiotic 4 capsules orally daily or 1 sachet orally daily for up to 5 weeks (starting between Day minus 7 to Day minus 4 and continuing through Day 28)
  Arms: Cohort II
Drug: Alclometasone cream — Topical alclometasone diproprionate cream 0.05% applied to face, hands, feet, neck, back and chest at bedtime for 4 weeks
  Arms: Cohort II

SUMMARY:
To assess the impact of prophylactic treatment on the incidence of adverse events in advanced NSCLC patients (post chemotherapy) treated with dacomitinib daily as a single agent. To assess the impact of an interrupted dacomitinib dosing schedule in Cycle 1 on the incidence of adverse events in first-line advanced NSCLC patients with an EGFR mutation (HER-1 mutation, HER-2 mutation or HER-2 amplification).

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non-Small Cell Lung Cancer (NSCLC).
* For Cohort I and Cohort II, advanced NSCLC patients must have received at least one prior regimen of systemic therapy which includes at least one standard chemotherapy for advanced NSCLC and who have failed (ie, progressed or intolerant due to toxicity which precludes further treatment) standard therapy for advanced or metastatic disease. To be considered intolerant to treatment, a patient must have received at least two cycles to be considered previously treated.
* For Cohort III, advanced NSCLC patients must not have received prior systemic treatment for their advanced disease and require a known EGFR (HER-1) mutation, HER-2 mutation or HER-2 amplification. Cohort III patients could have received prior adjuvant chemotherapy for Stage I-III disease or combined modality chemotherapy-radiation for Stage IIIA disease is allowed if treatment completed>12 months prior to enrollment.
* All cohorts, patients must have evidence of disease; however, measurable disease is not required to enroll.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Estimated creatinine clearance ≥15 mL/min.

Exclusion Criteria:

* Prior treatment with an EGFR-targeted or HER-targeted agent (all cohorts).
* Chemotherapy, radiotherapy, biological or investigational agents within 2 weeks of baseline disease assessments (all cohorts).
* Patients with known diffuse interstitial lung disease (all cohorts).
* Investigational therapy as only treatment for advanced NSCLC without administration of an approved chemotherapy for advanced NSCLC (for Cohort I and Cohort II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-12-26 (Actual); Primary Completion 2015-05-18 (Actual); Study Completion 2015-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (77):
- United States (75):
  - City of Hope, Duarte, California
  - St. Jude Heritage Healthcare, Fullerton, California
  - UCLA Hematology Oncology, Irvine, California
  - UC San Diego Medical Center - La Jolla, La Jolla, California
  - UC San Diego Moores Cancer Center - Investigational Drug Services, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Drug Management Only: UCLA West Medical Pharmacy, Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy Attn: Steven L. Wong, Pharm.D., Los Angeles, California
  - Drug Managment Only: UCLA West Medical Pharmacy, Los Angeles, California
  - Regulatory Management Only TRIO-US Central Administration, Los Angeles, California
  - Regulatory Management Only: TRIO-US Central Administration, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - Westwood Bowyer Clinic, Los Angeles, California
  - UCLA/Pasadena HealthCare, Pasadena, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - SANSUM Clinic, Santa Barbara, California
  - Cancer Center of Santa Barbara with SANSUM Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Hematology Oncology, Santa Monica, California
  - UCLA Santa Monica Medical Center & Orthopaedic Hospital, Santa Monica, California
  - Cancer Center of Santa Barbara with SANSUM Clinic, Solvang, California
  - City of Hope South Pasadena Cancer Center, South Pasadena, California
  - UCLA/Santa Clarita Valley Cancer Center, Valencia, California
  - UCLA Cancer Center, Westlake Village, California
  - Kaiser Permanente Colorado - Franklin, Denver, Colorado
  - St. Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Kaiser Permanente Colorado - Rock Creek, Lafayette, Colorado
  - Kaiser Permanente Colorado - Lonetree, Lonetree, Colorado
  - Michael and Dianne Bienes Comprehensive Cancer Center, Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Cancer Care of North Florida, PA, Lake City, Florida
  - Memorial West Cancer Institute, Pembroke Pines, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Summit Cancer Care,PC, Savannah, Georgia
  - Summit Cancer Care, PC, Savannah, Georgia
  - Rush University Medical Center, Division of Hematology & Oncology, Chicago, Illinois
  - Ships Drugs to: Emmanuel Semmes, RPh (or Ami Patel, Pharm D) University of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Josephine Ford Cancer Center-Downriver, Brownstown, Michigan
  - Henry Ford Medical Center - Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Henry Ford Hospital and Medical Center - West Bloomfield, West Bloomfield, Michigan
  - The West Clinic, PC, Corinth, Mississippi
  - The West Clinic, PC, Southaven, Mississippi
  - Mercy Clinic Cancer & Hematology-Branson, Branson, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Clinic Cancer and Hematology - Chub O-Reilly Cancer Center, Springfield, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Beth Israel Medical Center, New York, New York
  - Beth Israel Comprehensive Cancer Center, New York, New York
  - Columbia University Medical Center - The New York Presbyterian Hospital, New York, New York
  - Stony Brook University Medical Center-Cancer Center, Stony Brook, New York
  - Montefiore-Einstein Center for Cancer Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Oncology Specialists, PA, Hickory, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St Alexius Medical Center, Bismarck, North Dakota
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - The West Clinic, PC, Memphis, Tennessee
  - Investigational Product Center (IPC), Fort Worth, Texas
  - Investigational Products Center (IPC), Fort Worth, Texas
  - 'Fletcher Allen Health Care, Inc, Burlington, Vermont
  - Office of Clinical Trials Research, Fletcher Allen Health Care, Inc., Burlington, Vermont
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Cancer Institute - Issaquah, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471042&StudyName=Study%20Of%20Dacomitinib%20%28PF-00299804%29%20In%20Advanced%20NSCLC%20Patients%20%28Post%20Chemo%20Or%20Select%20First%20Line%29%20To%20Evaluate%20Prophylactic%20Interventio

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo): Open-label dacomitinib 45 milligram (mg) tablets orally (PO) taken once daily until progression of disease, intolerance to dacomitinib treatment, or participant withdrawal PLUS single-blind (participant blinded) doxycycline placebo capsules PO taken twice daily for 4 weeks (prophylactic treatment).
- Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg): Open-label dacomitinib 45 mg tablets PO taken once daily until progression of disease, intolerance to dacomitinib treatment, or participant withdrawal PLUS single-blind (participant blinded) doxycycline 100 mg capsules PO taken twice daily for 4 weeks (prophylactic treatment).
- Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate): Open-label dacomitinib 45 mg tablets PO taken once daily until progression of disease, intolerance to dacomitinib treatment, or participant withdrawal PLUS open-label topical alclometasone diproprionate cream 0.05 percent (%) applied to face, hands, feet, neck, back and chest at bedtime for 4 weeks (prophylactic treatment).
- Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone): Open-label dacomitinib 45 mg tablets PO taken once daily until progression of disease, intolerance to dacomitinib treatment, or participant withdrawal PLUS open-label VSL#3 probiotic 4 capsules PO taken once daily or 1 sachet PO taken once daily starting on either Days -7, -6, -5 or -4 per site/participant preference, and continuing through Cycle 1 Day 28 (for a total of up to 5 weeks [range of 32 to 35 days]) PLUS open-label topical alclometasone diproprionate cream 0.05% applied to face, hands, feet, neck, back and chest at bedtime for 4 weeks (prophylactic treatment).
- Cohort III (Dacomitinib 45 mg): Open-label dacomitinib 45 mg tablets PO, taken once daily Cycle 1 Day 1 through and including Cycle 1 Day 10; no dacomitinib was taken on Cycle 1 Days 11, 12, 13 and 14; resumption of dacomitinib 45 mg PO once daily taken continuously from Cycle 1 Day 15 onwards until progression of disease, intolerance to dacomitinib treatment, or participant withdrawal.
Period: Overall Study
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) | Cohort III (Dacomitinib 45 mg)
Started | 66 | 66 | 7 | 67 (An additional 5 participants were enrolled in Cohort II but not treated.) | 25
Completed | 33 | 42 | 7 | 38 | 13
Not Completed | 33 | 24 | 0 | 29 | 12
Not completed — Study terminated by sponsor | 1 | 0 | 0 | 1 | 7
Not completed — Withdrawal by Subject | 7 | 7 | 0 | 8 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Reason not specified | 9 | 4 | 0 | 10 | 2
Not completed — Death | 15 | 12 | 0 | 10 | 2

BASELINE CHARACTERISTICS:
Population: As Treated Population - included all participants who received at least 1 dose of study treatment assigned at enrollment.
Groups:
- Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo): Open-label dacomitinib 45 mg tablets PO taken once daily until progression of disease, intolerance to dacomitinib treatment, or participant withdrawal PLUS single-blind (participant blinded) doxycycline placebo capsules PO taken twice daily for 4 weeks (prophylactic treatment).
- Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate): Open-label dacomitinib 45 mg tablets PO taken once daily until progression of disease, intolerance to dacomitinib treatment, or participant withdrawal PLUS open-label topical alclometasone diproprionate cream 0.05% applied to face, hands, feet, neck, back and chest at bedtime for 4 weeks (prophylactic treatment).
- Total: Total of all reporting groups
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) | Cohort III (Dacomitinib 45 mg) | Total
Number analyzed (Participants) | 66 | 66 | 7 | 67 | 25 | 231
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (10.38) | 64.4 (10.55) | 61.3 (7.67) | 66.0 (9.63) | 64.2 (14.29) | 64.9 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 27 | 2 | 24 | 18 | 109
  Male | 28 | 39 | 5 | 43 | 7 | 122

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Select Dermatologic Adverse Events of Interest (SDAEI) (All Causality, All Grade) in the First 8 Weeks of Treatment by Treatment Arm for Cohort I
Description: SDAEI of all causality and all grades were evaluated in participants in Cohort I. These SDAEIs included dermatitis acneiform, dry skin, exfoliative rash, nail discoloration, nail disorder, paronychia, pruritus, rash, skin exfoliation, skin fissures, skin infection, skin laceration and skin ulcer.
  95% confidence interval (CI) calculated using exact method based on binomial distribution.
  After protocol amendment 1, Arm C was removed from Cohort I and enrollment to Arm C was terminated. Only 7 participants were enrolled in Cohort I Arm C as a result. Given the smaller sample size, analyse of Outcome Measure 1 was not conducted in Cohort I Arm C.
Time Frame: First 8 Weeks of Treatment
Population: Evaluable Population - included all participants who received the study treatment assigned at enrollment, but did not discontinue dacomitinib treatment less than 6 weeks from first dosing due to either disease progression or death.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg)
Number analyzed (Participants) | 58 | 56
Percentage of Participants | 79.3 [66.6 to 88.8] | 75.0 [61.6 to 85.6]

2. Primary Outcome: Percentage of Participants With SDAEI (All Causality, Grade Greater Than or Equal to [≥] 2) in the First 8 Weeks of Treatment by Treatment Arm for Cohort I
Description: SDAEI of all causality and Grade ≥2 were evaluated in participants in Cohort I. These SDAEIs included dermatitis acneiform, dry skin, exfoliative rash, nail discoloration, nail disorder, paronychia, pruritus, rash, skin exfoliation, skin fissures, skin infection, skin laceration and skin ulcer. Adverse events (AEs) were graded for severity using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, Version 4.0).
  95% CI calculated using exact method based on binomial distribution. After protocol amendment 1, Arm C was removed from Cohort I and enrollment to Arm C was terminated. Only 7 participants were enrolled in Cohort I Arm C as a result. Given the smaller sample size, analyse of Outcome Measure 2 was not conducted in Cohort I Arm C.
Time Frame: First 8 Weeks of Treatment
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg)
Number analyzed (Participants) | 58 | 56
Percentage of Participants | 46.6 [33.3 to 60.1] | 23.2 [13.0 to 36.4]

3. Primary Outcome: Mean Change From Baseline (Cycle 1 Day 1) Skindex-16 Scale Scores (Total Score, Symptoms Score, Emotion Score, and Functioning Score) by Treatment Arm for Cohort I
Description: Patient Reported Outcomes (PROs) of Health Related Quality of Life (HRQoL) & disease/treatment-related symptoms were assessed using Dermatologic Survey (Skindex-16) that assesses "bother". It includes 3 multi-item scales: symptoms, emotions & functioning. Individual scaled scores & total scores were determined. Skindex questions were transformed to a linear scale of 0 (never bothered) to 100 (always bothered). Subscale scores are an average of non-missing questions in a given scale if greater than (>) 75% of total subscale questions are non-missing. The Total Score is an average of all non-missing questions in the Skindex if >75% of total questions are non-missing. A negative change score represents a better quality of life. A change score of 10 points is considered clinically significant.
  Skindex completion criteria were defined as completion of 3 out of 4 items for questions 1 to 4, 6 out of 7 items for questions 5 to 11, 4 out of 5 items for questions 12 to 16 for the visit.
Time Frame: First 8 Weeks of Treatment
Population: PRO Skindex Analysis Population: participants that met primary endpoint analysis & Skindex specific criteria: a) Skindex completion criteria (as above) for initial visit & end of Cycle 2 or EoT visit; b) Skindex completion criteria for at least 5 of 6 visits between initial visit & end of Cycle 2 visit. n = number of participants completing scale.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate)
Number analyzed (Participants) | 42 | 42 | 4
Score on a scale
  Symptoms: Cycle 1 Day 8 (n=41, 42, 4) | 2.3 (10.12) | -1.1 (10.91) | 9.4 (14.18)
  Symptoms: Cycle 1 Day 15 (n=41, 42, 3) | 21.4 (30.98) | 5.0 (19.82) | 30.6 (42.56)
  Symptoms: Cycle 1 Day 22 (n=42, 40, 4) | 18.0 (25.76) | 6.8 (20.45) | 32.3 (25.54)
  Symptoms: Cycle 2 Day 1 (n=41, 42, 4) | 14.7 (23.74) | 6.3 (15.38) | 14.6 (18.48)
  Symptoms: Cycle 2 Day 8 (n=42, 39, 4) | 17.8 (26.78) | 9.8 (20.00) | 13.5 (19.36)
  Symptoms: Cycle 2 Day 15 (n=37, 40, 4) | 16.6 (21.10) | 9.2 (19.54) | 19.8 (28.74)
  Symptoms: Cycle 2 Day 22 (n=35, 39, 4) | 15.4 (22.34) | 12.9 (22.72) | 14.6 (15.40)
  Symptoms: EoT (n=7, 3, 0) | 13.1 (32.85) | 16.7 (19.09) | NA (NA) — NA = not applicable. The number of participants completing the scale at this timepoint was 0.
  Emotion: Cycle 1 Day 8 (n=41, 42, 4) | 3.7 (21.08) | -2.5 (12.11) | 7.3 (14.68)
  Emotion: Cycle 1 Day 15 (n=41, 42, 3) | 20.7 (28.51) | 2.9 (17.14) | 29.8 (45.03)
  Emotion: Cycle 1 Day 22 (n=42, 40, 4) | 17.7 (27.67) | 3.7 (16.07) | 37.7 (32.44)
  Emotion: Cycle 2 Day 1 (n=41, 42, 4) | 15.6 (25.15) | 6.5 (15.25) | 23.4 (30.15)
  Emotion: Cycle 2 Day 8 (n=42, 39, 4) | 15.1 (25.55) | 6.3 (17.28) | 21.6 (35.76)
  Emotion: Cycle 2 Day 15 (n=37, 40, 4) | 13.0 (22.70) | 8.4 (20.20) | 21.0 (40.49)
  Emotion: Cycle 2 Day 22 (n=35, 39, 4) | 14.8 (25.91) | 12.0 (23.73) | 10.9 (17.39)
  Emotion: EoT (n=7, 3, 0) | 9.9 (21.27) | 22.2 (21.34) | NA (NA) — The number of participants completing the scale at this timepoint was 0.
  Functioning: Cycle 1 Day 8 (n=41, 42, 4) | 3.1 (17.60) | -1.2 (5.50) | -0.8 (1.67)
  Functioning: Cycle 1 Day 15 (n=41, 42, 3) | 11.1 (21.41) | 0.6 (7.47) | 24.4 (42.34)
  Functioning: Cycle 1 Day 22 (n=42, 40, 4) | 11.7 (21.68) | 1.9 (8.86) | 33.3 (31.39)
  Functioning: Cycle 2 Day 1 (n=41, 42, 4) | 8.5 (21.53) | 2.1 (7.72) | 20.0 (21.26)
  Functioning: Cycle 2 Day 8 (n=42, 39, 4) | 7.0 (18.51) | 2.4 (9.52) | 12.5 (20.79)
  Functioning: Cycle 2 Day 15 (n=37, 40, 4) | 8.3 (22.20) | 2.7 (10.58) | 13.3 (22.44)
  Functioning: Cycle 2 Day 22 (n=35, 39, 4) | 7.8 (22.32) | 5.4 (13.78) | 14.2 (20.44)
  Functioning: EoT (n=7, 3, 0) | 8.6 (11.84) | 14.4 (25.02) | NA (NA) — The number of participants completing the scale at this timepoint was 0.
  Total: Cycle 1 Day 8 (n=41, 42, 4) | 3.2 (15.91) | -1.7 (8.07) | 5.3 (9.36)
  Total: Cycle 1 Day 15 (n=41, 42, 3) | 17.9 (25.09) | 2.7 (13.08) | 28.4 (43.52)
  Total: Cycle 1 Day 22 (n=42, 40, 4) | 15.9 (23.39) | 4.0 (13.33) | 35.0 (29.97)
  Total: Cycle 2 Day 1 (n=41, 42, 4) | 13.1 (20.74) | 5.1 (11.65) | 20.2 (21.75)
  Total: Cycle 2 Day 8 (n=42, 39, 4) | 13.2 (21.17) | 6.0 (13.49) | 16.8 (24.54)
  Total: Cycle 2 Day 15 (n=37, 40, 4) | 12.4 (20.39) | 6.8 (14.84) | 18.4 (31.50)
  Total: Cycle 2 Day 22 (n=35, 39, 4) | 12.7 (21.24) | 10.1 (18.36) | 12.9 (17.22)
  Total: EoT (n=7, 3, 0) | 10.3 (18.79) | 18.4 (18.64) | NA (NA) — The number of participants completing the scale at this timepoint was 0.

4. Primary Outcome: Percentage of Participants With Diarrhea AEs (All Causality, All Grade and Grade ≥2) in the First 8 Weeks of Treatment for Cohort II
Description: Diarrhea AEs of all causality, all grade and Grade ≥2 were evaluated in participants in Cohort II. AEs were graded for severity using the NCI-CTCAE, Version 4.0.
  95% CI calculated using exact method based on binomial distribution.
Time Frame: First 8 Weeks of Treatment
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone)
Number analyzed (Participants) | 59
Percentage of Participants
  All Causality, All Grade | 83.1 [71.0 to 91.6]
  All Causality, Grade ≥2 | 39.0 [26.5 to 52.6]

5. Primary Outcome: Mean Change From Baseline (Cycle 1 Day 1) Modified Oral Mucositis Daily Questionnaire (OMDQ) Scores (Mouth and Throat Soreness Categories and Scale, and Diarrhea Categories and Scale) for Cohort II
Description: Diarrhea severity was assessed using the modified-OMDQ. This questionnaire is comprised of 6 questions in total; however, only two items relate to diarrhea symptoms (item 5 and item 6). Symptoms scores were developed for both the full questionnaire and for the diarrhea-only questions for each completed survey. Mucositis questions were transformed to a score range of 0 to 10. Increasing OMDQ values are associated with greater symptom burden.
  Modified OMDQ completion criteria were defined as completion of all 4 questions (questions 2, 4, 5 and 6).
  M/T = mouth and throat.
Time Frame: Cycles 1, 2, 3, 4, 5, and 6, EoT and Follow-up
Population: PRO Modified OMDQ Analysis Population; participants meeting primary endpoint analysis & modified OMDQ specific criteria: a) Modified OMDQ completion criteria for initial visit & end of Cycle 2 or EoT visit; b) Completion criteria for at least 5 of 6 visits between initial & end of Cycle 2 visit. n = number of participants completing scale.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone)
Number analyzed (Participants) | 37
Score on a scale
  M/T Soreness Categories: Cycle 1 Day 8 (n=37) | 0.8 (2.05)
  M/T Soreness Categories: Cycle 1 Day 15 (n=37) | 2.5 (3.12)
  M/T Soreness Categories: Cycle 1 Day 22 (n=37) | 2.6 (2.97)
  M/T Soreness Categories: Cycle 2 Day 1 (n=37) | 2.5 (2.43)
  M/T Soreness Categories: Cycle 2 Day 8 (n=35) | 1.9 (2.30)
  M/T Soreness Categories: Cycle 2 Day 15 (n=36) | 1.7 (1.97)
  M/T Soreness Categories: Cycle 2 Day 22 (n=27) | 1.6 (1.85)
  M/T Soreness Categories: Cycle 3 Day 1 (n=19) | 2.1 (2.09)
  M/T Soreness Categories: Cycle 4 Day 1 (n=13) | 1.7 (2.14)
  M/T Soreness Categories: Cycle 5 Day 1 (n=10) | 1.0 (1.29)
  M/T Soreness Categories: Cycle 6 Day 1 (n=8) | 0.3 (0.88)
  M/T Soreness Categories: EoT (n=30) | 1.4 (2.34)
  M/T Soreness Categories: Follow-up (n=22) | 0.3 (2.48)
  M/T Soreness Scale: Cycle 1 Day 8 (n=37) | 1.0 (2.00)
  M/T Soreness Scale: Cycle 1 Day 15 (n=37) | 2.5 (3.00)
  M/T Soreness Scale: Cycle 1 Day 22 (n=37) | 2.2 (2.51)
  M/T Soreness Scale: Cycle 2 Day 1 (n=37) | 2.2 (2.28)
  M/T Soreness Scale: Cycle 2 Day 8 (n=35) | 1.7 (1.97)
  M/T Soreness Scale: Cycle 2 Day 15 (n=36) | 1.6 (1.83)
  M/T Soreness Scale: Cycle 2 Day 22 (n=27) | 1.9 (2.45)
  M/T Soreness Scale: Cycle 3 Day 1 (n=19) | 2.2 (2.81)
  M/T Soreness Scale: Cycle 4 Day 1 (n=13) | 1.6 (2.81)
  M/T Soreness Scale: Cycle 5 Day 1 (n=10) | 1.0 (1.76)
  M/T Soreness Scale: Cycle 6 Day 1 (n=8) | 0.1 (0.35)
  M/T Soreness Scale: EoT (n=30) | 1.3 (1.78)
  M/T Soreness Scale: Follow-up (n=22) | 0.5 (1.68)
  Diarrhea Categories: Cycle 1 Day 8 (n=37) | 2.1 (2.67)
  Diarrhea Categories: Cycle 1 Day 15 (n=37) | 3.2 (2.94)
  Diarrhea Categories: Cycle 1 Day 22 (n=36) | 3.9 (3.19)
  Diarrhea Categories: Cycle 2 Day 1 (n=37) | 3.0 (2.83)
  Diarrhea Categories: Cycle 2 Day 8 (n=34) | 2.2 (3.00)
  Diarrhea Categories: Cycle 2 Day 15 (n=36) | 2.1 (3.13)
  Diarrhea Categories: Cycle 2 Day 22 (n=27) | 2.7 (3.10)
  Diarrhea Categories: Cycle 3 Day 1 (n=19) | 2.8 (2.75)
  Diarrhea Categories: Cycle 4 Day 1 (n=13) | 2.3 (3.14)
  Diarrhea Categories: Cycle 5 Day 1 (n=10) | 3.8 (3.39)
  Diarrhea Categories: Cycle 6 Day 1 (n=8) | 1.9 (2.22)
  Diarrhea Categories: EoT (n=30) | 1.9 (3.39)
  Diarrhea Categories: Follow-up (n=22) | -0.1 (0.94)
  Diarrhea Scale: Cycle 1 Day 8 (n=37) | 1.2 (1.89)
  Diarrhea Scale: Cycle 1 Day 15 (n=37) | 2.4 (2.55)
  Diarrhea Scale: Cycle 1 Day 22 (n=36) | 3.0 (2.96)
  Diarrhea Scale: Cycle 2 Day 1 (n=37) | 2.5 (2.61)
  Diarrhea Scale: Cycle 2 Day 8 (n=34) | 2.0 (2.75)
  Diarrhea Scale: Cycle 2 Day 15 (n=35) | 1.7 (2.71)
  Diarrhea Scale: Cycle 2 Day 22 (n=27) | 2.0 (2.16)
  Diarrhea Scale: Cycle 3 Day 1 (n=19) | 2.4 (2.34)
  Diarrhea Scale: Cycle 4 Day 1 (n=13) | 1.8 (2.13)
  Diarrhea Scale: Cycle 5 Day 1 (n=10) | 2.7 (2.31)
  Diarrhea Scale: Cycle 6 Day 1 (n=8) | 1.5 (1.93)
  Diarrhea Scale: EoT (n=30) | 1.6 (2.87)
  Diarrhea Scale: Follow-up (n=22) | -0.1 (0.71)

6. Primary Outcome: Percentage of Participants With SDAEI (All Causality, All Grade) in the First 8 Weeks of Treatment for Cohort II
Description: SDAEI of all causality and all grades were evaluated in participants in Cohort II. These SDAEIs included dermatitis acneiform, dry skin, exfoliative rash, nail discoloration, nail disorder, paronychia, pruritus, rash, skin exfoliation, skin fissures, skin infection, skin laceration and skin ulcer.
  95% CI calculated using exact method based on binomial distribution.
Time Frame: First 8 Weeks of Treatment
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone)
Number analyzed (Participants) | 59
Percentage of Participants | 79.7 [67.2 to 89.0]

7. Primary Outcome: Percentage of Participants With SDAEI (All Causality, Grade ≥2) in the First 8 Weeks of Treatment for Cohort II
Description: SDAEI of all causality and Grade ≥2 were evaluated in participants in Cohort II. These SDAEIs included dermatitis acneiform, dry skin, exfoliative rash, nail discoloration, nail disorder, paronychia, pruritus, rash, skin exfoliation, skin fissures, skin infection, skin laceration and skin ulcer. AEs were graded for severity using the NCI-CTCAE, Version 4.0.
  95% CI calculated using exact method based on binomial distribution.
Time Frame: First 8 Weeks of Treatment
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone)
Number analyzed (Participants) | 59
Percentage of Participants | 35.6 [23.6 to 49.1]

8. Primary Outcome: Mean Change From Baseline (Cycle 1 Day 1) Skindex-16 Scale Scores (Total Score, Symptoms Score, Emotion Score, and Functioning Score) for Cohort II
Description: PROs of HRQoL and disease/treatment-related symptoms were assessed using Dermatologic Survey (Skindex-16) that assesses "bother". It includes 3 multi-item scales: symptoms, emotions & functioning. Individual scaled scores & total scores were determined. Skindex questions were transformed to a linear scale of 0 (never bothered) to 100 (always bothered). Subscale scores are an average of non-missing questions in a given scale if > 75% of total subscale questions are non-missing. The Total Score is an average of all non-missing questions in the Skindex if >75% of total questions are non-missing. A negative change score represents a better quality of life. A change score of 10 points is considered clinically significant.
  Skindex completion criteria were defined as completion of 3 out of 4 items for questions 1 to 4, 6 out of 7 items for questions 5 to 11, 4 out of 5 items for questions 12 to 16 for the visit.
Time Frame: Cycles 1, 2, 3, 4, 5, and 6, EoT and Follow-up
Population: PRO Skindex Analysis Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone)
Number analyzed (Participants) | 40
Score on a scale
  Symptoms: Cycle 1 Day 8 (n=40) | 0.1 (8.31)
  Symptoms: Cycle 1 Day 15 (n=40) | 11.4 (21.25)
  Symptoms: Cycle 1 Day 22 (n=40) | 11.4 (18.17)
  Symptoms: Cycle 2 Day 1 (n=40) | 11.4 (19.84)
  Symptoms: Cycle 2 Day 8 (n=38) | 13.5 (20.88)
  Symptoms: Cycle 2 Day 15 (n=38) | 14.7 (17.83)
  Symptoms: Cycle 2 Day 22 (n=30) | 13.6 (16.30)
  Symptoms: Cycle 3 Day 1 (n=21) | 12.7 (19.56)
  Symptoms: Cycle 4 Day 1 (n=15) | 11.9 (18.69)
  Symptoms: Cycle 5 Day 1 (n=11) | 8.0 (22.24)
  Symptoms: Cycle 6 Day 1 (n=8) | 12.0 (32.15)
  Symptoms: EoT (n=33) | 10.4 (21.33)
  Symptoms: Follow-up (n=23) | 7.1 (23.15)
  Emotion: Cycle 1 Day 8 (n=40) | 1.0 (11.79)
  Emotion: Cycle 1 Day 15 (n=40) | 8.7 (23.57)
  Emotion: Cycle 1 Day 22 (n=40) | 12.3 (24.63)
  Emotion: Cycle 2 Day 1 (n=40) | 10.2 (21.36)
  Emotion: Cycle 2 Day 8 (n=38) | 10.3 (21.77)
  Emotion: Cycle 2 Day 15 (n=37) | 13.5 (17.10)
  Emotion: Cycle 2 Day 22 (n= 30) | 12.6 (19.86)
  Emotion: Cycle 3 Day 1 (n=21) | 11.0 (17.97)
  Emotion: Cycle 4 Day 1 (n=14) | 11.5 (14.65)
  Emotion: Cycle 5 Day 1 (n=11) | 7.8 (21.43)
  Emotion: Cycle 6 Day 1 (n=8) | 6.8 (22.67)
  Emotion: EoT (n=33) | 8.5 (23.38)
  Emotion: Follow-up (n=23) | 7.1 (22.74)
  Functioning: Cycle 1 Day 8 (n=40) | 0.5 (3.58)
  Functioning: Cycle 1 Day 15 (n=40) | 4.3 (13.34)
  Functioning: Cycle 1 Day 22 (n=40) | 8.8 (17.55)
  Functioning: Cycle 2 Day 1 (n=40) | 7.3 (15.25)
  Functioning: Cycle 2 Day 8 (n=38) | 6.2 (15.33)
  Functioning: Cycle 2 Day 15 (n=38) | 7.0 (11.75)
  Functioning: Cycle 2 Day 22 (n=30) | 7.2 (10.06)
  Functioning: Cycle 3 Day 1 (n=21) | 5.9 (8.09)
  Functioning: Cycle 4 Day 1 (n=15) | 6.9 (10.12)
  Functioning: Cycle 5 Day 1 (n=11) | 5.5 (12.93)
  Functioning: Cycle 6 Day 1 (n=8) | 7.1 (15.58)
  Functioning: EoT (n=33) | 7.7 (17.35)
  Functioning: Follow-up (n=23) | 5.4 (18.55)
  Total: Cycle 1 Day 8 (n=40) | 0.6 (6.83)
  Total: Cycle 1 Day 15 (n=40) | 8.0 (18.73)
  Total: Cycle 1 Day 22 (n=40) | 11.0 (19.59)
  Total: Cycle 2 Day 1 (n=40) | 9.6 (17.38)
  Total: Cycle 2 Day 8 (n=38) | 9.9 (17.79)
  Total: Cycle 2 Day 15 (n=38) | 11.8 (14.13)
  Total: Cycle 2 Day 22 (n=30) | 11.2 (14.14)
  Total: Cycle 3 Day 1 (n=21) | 9.8 (14.11)
  Total: Cycle 4 Day 1 (n=15) | 10.2 (12.49)
  Total: Cycle 5 Day 1 (n=11) | 7.1 (18.60)
  Total: Cycle 6 Day 1 (n=8) | 8.2 (22.43)
  Total: EoT (n=33) | 8.7 (19.74)
  Total: Follow-up (n=23) | 6.6 (20.52)

9. Secondary Outcome: Percentage of Participants Receiving Any Concomitant Drug or Non-Drug Treatment for SDAEI, Diarrhea and Mucositis for Cohort I by Treatment Arm, Cohort II, and Cohort III
Description: Medications used concomitantly for SDAEIs, diarrhea and mucositis were evaluated for all participants who received dacomitinib on a continuous basis with a preemptive prophylactic (Cohorts I and II) or as an interrupted dosing regimen (Cohort III).
Time Frame: Screening to the Post-Teatment Follow-Up Visit (at least 28 days and no more than 35 days after the end of dacomitinib treatment due to progression of disease, intolerance to dacomitinib treatment, or participant withdrawal)
Population: As Treated Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) | Cohort III (Dacomitinib 45 mg)
Number analyzed (Participants) | 66 | 66 | 7 | 67 | 25
Percentage of Participants
  Any Concomitant Drug | 69.7 | 60.6 | 85.7 | 82.1 | 88.0
  Any Non-Drug Treatment | 16.7 | 16.7 | 42.9 | 20.9 | 44.0

10. Primary Outcome: Mean Area Under the Plasma Concentration Time Curve From 0 to 24 Hours (AUC0-24) and From 0 to 120 Hours (AUC0-120) for Dacomitinib and Its Metabolite PF-05199265 on Cycle 1 Days 10 to 15 for Cohort III
Description: AUC0-24 is the area under the plasma concentration-time curve (AUC) from time 0 to 24 hours post-dose. AUC0-120 is the AUC from time 0 to 120 hours post-dose. AUC was calculated by the linear trapezoidal method using a non-compartmental pharmacokinetic (PK) analysis.
  ng*hr/mL = nanogram hours per milliliter
Time Frame: Cycle 1 Day 10: Pre-dose and 2, 4, 6, 24, 48, 72, 96, and 120 hours post-dose (the 120 hour sample was obtained on Day 15 pre-dose).
Population: Dose-Compliant participants only. Participants were considered dose-compliant when they received all planned doses at the same dose level right before sample collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort III (Dacomitinib 45 mg)
Number analyzed (Participants) | 23
ng*hr/mL
  Dacomitinib AUC0-24 | 1712.88 (35)
  Dacomitinib AUC0-120 | 5743.60 (32)
  PF-05199265 AUC0-24 | 184.62 (139)
  PF-05199265 AUC0-120 | 742.32 (129)

11. Primary Outcome: Mean Maximum Observed Plasma Concentrations (Cmax) for Dacomitinib and Its Metabolite PF-05199265 on Cycle 1 Days 10 to 15 for Cohort III
Description: Cmax was obtained from direct inspection of the data. ng/mL = nanograms per milliliter
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort III (Dacomitinib 45 mg)
Number analyzed (Participants) | 23
ng/mL
  Dacomitinib Cmax | 79.68 (36)
  PF-05199265 Cmax | 8.5176 (137)

12. Primary Outcome: Median Time of Occurrence of Cmax (Tmax) for Dacomitinib and Its Metabolite PF-05199265 on Cycle 1 Days 10 to 15 for Cohort III
Description: Tmax was obtained from direct inspection of the data as the time of first occurence of Cmax.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Cohort III (Dacomitinib 45 mg)
Number analyzed (Participants) | 23
hours (hr)
  Dacomitinib Tmax | 5.850 (53) [0 to 24.30]
  PF-05199265 Tmax | 5.980 (126) [0 to 24.30]

13. Secondary Outcome: Mean AUC From 0 to the End of the Dosing Interval (AUC0-tau) for Dacomitinib and Its Metabolite PF-05199265 on Cycle 2 Day 1 for Cohort I
Description: AUCtau was the AUC from time 0 to the end of the dosing interval, where the dosing interval was 24 hours. AUCtau was calculated by the linear/log trapezoidal method using a non-compartmental PK analysis.
Time Frame: Cycle 2 Day 1: pre-dose and at 2, 4, 6, and 24 hours post-dose
Population: Dose-Compliant participants only. Participants were considered dose-compliant when they received at least 14 consecutive doses at the same dose level right before sample collection.
  Number of participants analyzed is the number of participants contributing to the summary statistics.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate)
Number analyzed (Participants) | 27 | 27 | 2
ng*hr/mL
  Dacomitinib AUC0-tau | 1801.96 (59) | 1869.23 (37) | 1412.42 (63)
  PF-05199265 AUC0-tau | 164.520 (89) | 112.306 (139) | 366.933 (107)

14. Secondary Outcome: Mean Cmax for Dacomitinib and Its Metabolite PF-05199265 on Cycle 2 Day 1 for Cohort I
Description: Cmax was obtained from direct inspection of the data.
Time Frame: Cycle 2 Day 1: pre-dose and at 2, 4, 6, and 24 hours post-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate)
Number analyzed (Participants) | 31 | 27 | 3
ng/mL
  Dacomitinib Cmax | 88.15 (57) | 89.79 (36) | 98.08 (89)
  PF-05199265 Cmax | 7.7426 (80) | 5.2901 (141) | 8.8545 (260)

15. Secondary Outcome: Median Tmax for Dacomitinib and Its Metabolite PF-05199265 on Cycle 2 Day 1 for Cohort I
Description: Tmax was obtained from direct inspection of the data as the time of first occurence of Cmax.
Time Frame: Cycle 2 Day 1: pre-dose and at 2, 4, 6, and 24 hours post-dose
Population: as for outcome 13
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate)
Number analyzed (Participants) | 31 | 27 | 3
hr
  Dacomitinib Tmax | 4.000 (67) [0 to 24.00] | 6.000 (67) [0 to 24.30] | 6.580 (108) [4.02 to 22.20]
  PF-05199265 Tmax | 4.050 (82) [0 to 24.10] | 4.020 (125) [0 to 24.30] | 6.580 (105) [0 to 22.20]

16. Secondary Outcome: Mean Apparent Clearance (CL/F) for Dacomitinib on Cycle 2 Day 1 for Cohort I
Description: CL/F was calculated as dose/AUCtau.
Time Frame: Cycle 2 Day 1: pre-dose and at 2, 4, 6, and 24 hours post-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate)
Number analyzed (Participants) | 31 | 27 | 3
Liters per hour | 29.94 (85) | 24.07 (37) | 34.24 (45)

17. Secondary Outcome: Mean Plasma Trough Concentrations (Ctrough) for Dacomitinib by Visit for Cohorts I, II and III
Description: Ctrough was the pre-dose plasma concentration of dacomitinib at steady state obtained from direct inspection of the data.
  Number of participants analyzed is the total number of participants in the treatment group in the indicated population, n is the number of participants contributing to the summary statistics.
Time Frame: Cohorts I to III: Pre-dose on Day 1 of Cycle 3 to 10.
Population: Dose-Compliant participants only. Participants were considered dose-compliant when they received at least 14 consecutive doses at the same dose level right before sample collection in Cohorts I, II and III.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) | Cohort III (Dacomitinib 45 mg)
Number analyzed (Participants) | 34 | 32 | 5 | 15 | 23
ng/mL
  Cycle 3 Day 1 (n=13, 15, 3, 14, 15) | 65.477 (50) | 65.063 (55) | 56.212 (46) | 66.338 (58) | 55.780 (40)
  Cycle 4 Day 1 (n=8, 7, 2, 5, 13) | 61.592 (36) | 67.109 (29) | 65.466 (49) | 71.116 (49) | 55.644 (42)
  Cycle 5 Day 1 (n=3, 6, 2, 3, 12) | 89.970 (38) | 68.012 (39) | 69.649 (63) | 66.082 (33) | 53.116 (44)
  Cycle 6 Day 1 (n=2, 5, 1, 2, 10) | 15.578 (1208) | 72.856 (47) | 46.000 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 9.201 (3760) | 52.603 (52)
  Cycle 7 Day 1 (n=2, 1, 1, 1, 8) | 59.086 (47) | 40.900 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 59.900 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 42.600 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 55.685 (21)
  Cycle 8 Day 1 (n=2, 2, 1, 2, 8) | 61.430 (90) | 58.988 (31) | 47.00 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 64.296 (35) | 51.559 (24)
  Cycle 9 Day 1 (n=2, 2, 1, 2, 6) | 64.747 (72) | 58.928 (31) | 46.000 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 64.115 (30) | 44.865 (50)
  Cycle 10 Day 1 (n=1, 2, 1, 2, 4) | 51.400 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 54.041 (48) | 58.800 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 71.695 (26) | 55.362 (32)

18. Secondary Outcome: Mean Plasma Ctrough for PF-05199265 by Visit for Cohorts I, II and III
Description: Ctrough was the pre-dose plasma concentration of the dacomitinib metabolite PF-05199265 at steady state obtained from direct inspection of the data.
  Number of participants analyzed is the total number of participants in the treatment group in the indicated population, n is the number of participants contributing to the summary statistics.
Time Frame: Cohorts I to III: Pre-dose on Day 1 of Cycle 3 to 10.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) | Cohort III (Dacomitinib 45 mg)
Number analyzed (Participants) | 34 | 32 | 5 | 15 | 23
ng/mL
  Cycle 3 Day 1 (n=13, 15, 3, 14, 15) | 6.988 (60) | 4.653 (133) | 10.220 (11) | 7.814 (59) | 9.967 (149)
  Cycle 4 Day 1 (n=8, 7, 2, 5, 13) | 5.555 (71) | 5.271 (242) | 8.522 (15) | 6.848 (82) | 11.759 (113)
  Cycle 5 Day 1 (n=3, 6, 2, 3, 12) | 4.356 (55) | 4.989 (58) | 8.522 (10) | 5.850 (115) | 10.510 (124)
  Cycle 6 Day 1 (n=2, 5, 1, 2, 10) | 5.020 (70) | 6.523 (123) | 8.150 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 1.261 (937) | 7.844 (125)
  Cycle 7 Day 1 (n=2, 1, 1, 1, 8) | 4.850 (49) | 23.900 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 8.560 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 6.680 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 8.203 (105)
  Cycle 8 Day 1 (n=2, 2, 1, 2, 8) | 5.349 (54) | 6.085 (476) | 10.100 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 10.844 (38) | 8.205 (117)
  Cycle 9 Day 1 (n=2, 2, 1, 2, 6) | 4.271 (34) | 6.448 (612) | 9.720 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 9.159 (58) | 6.963 (88)
  Cycle 10 Day 1 (n=1, 2, 1, 2, 4) | 3.460 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 6.892 (305) | 10.700 (NA) — Geometric mean coefficient of variation is not calculable as n=1. | 9.442 (26) | 6.364 (154)

ADVERSE EVENTS:
Time Frame: Reported AEs and serious AEs (SAEs) included events starting from the time participant had taken at least 1 dose of study drug through and including 28 calendar days after the last dose of study drug, with a median of 12 weeks.
Description: The same event may appear as both an AE & SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant & non-serious in another, or 1 participant may have experienced both a serious & non-serious event during the study. Summaries inclusive of events occurring after start of treatment.
Arm/Group | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) | Cohort III (Dacomitinib 45 mg)
Serious Adverse Events (participants affected / at risk) | 25/66 | 27/66 | 3/7 | 22/67 | 6/25
Other Adverse Events (participants affected / at risk) | 65/66 | 66/66 | 7/7 | 64/67 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) (N=66) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) (N=66) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) (N=7) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) (N=67) | Cohort III (Dacomitinib 45 mg) (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 1
Asthenia (General disorders) | 2 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 7 | 7 | 0 | 8 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 2 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 5 | 1
Septic shock (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 3 | 0 | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort I: Arm A (Dacomitinib 45 mg + Doxycycline Placebo) (N=66) | Cohort I: Arm B (Dacomitinib 45 mg + Doxycycline 100 mg) (N=66) | Cohort I: Arm C (Dacomitinib 45mg+Alclometasone Diproprionate) (N=7) | Cohort II (Dacomitinib 45mg + VSL#3 Probiotic + Alclometasone) (N=67) | Cohort III (Dacomitinib 45 mg) (N=25)
Anaemia (Blood and lymphatic system disorders) | 10 | 7 | 3 | 5 | 3
Tachycardia (Cardiac disorders) | 1 | 4 | 0 | 3 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 5 | 4 | 0 | 2 | 3
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 2
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0 | 1 | 2
Vision blurred (Eye disorders) | 0 | 1 | 2 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 7 | 7 | 0 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3 | 0 | 2 | 2
Cheilitis (Gastrointestinal disorders) | 3 | 1 | 1 | 3 | 1
Constipation (Gastrointestinal disorders) | 9 | 14 | 2 | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 54 | 52 | 7 | 54 | 23
Dry mouth (Gastrointestinal disorders) | 4 | 5 | 1 | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 10 | 0 | 2 | 3
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 4 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 28 | 31 | 2 | 20 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0
Oral pain (Gastrointestinal disorders) | 2 | 4 | 0 | 7 | 2
Stomatitis (Gastrointestinal disorders) | 10 | 12 | 3 | 14 | 16
Vomiting (Gastrointestinal disorders) | 16 | 23 | 3 | 14 | 5
Asthenia (General disorders) | 4 | 7 | 2 | 3 | 1
Chest discomfort (General disorders) | 2 | 1 | 0 | 0 | 2
Chills (General disorders) | 5 | 0 | 4 | 1 | 1
Fatigue (General disorders) | 24 | 27 | 3 | 20 | 5
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 4
Malaise (General disorders) | 0 | 2 | 1 | 1 | 0
Mucosal inflammation (General disorders) | 19 | 21 | 2 | 12 | 5
Oedema peripheral (General disorders) | 6 | 4 | 1 | 4 | 3
Pain (General disorders) | 5 | 7 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 4 | 1 | 0 | 4
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Immunosuppression (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 2 | 0 | 4 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 1 | 0 | 2
Mucosal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 12 | 10 | 3 | 9 | 16
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 2 | 2
Rash pustular (Infections and infestations) | 4 | 2 | 0 | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 3 | 7
Urinary tract infection (Infections and infestations) | 8 | 7 | 1 | 2 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 5 | 0 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 2 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 6 | 1 | 1 | 3 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 1 | 0 | 4 | 1
Blood creatinine increased (Investigations) | 8 | 5 | 1 | 3 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 15 | 15 | 2 | 8 | 7
Decreased appetite (Metabolism and nutrition disorders) | 24 | 22 | 3 | 25 | 14
Dehydration (Metabolism and nutrition disorders) | 15 | 15 | 1 | 9 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 1 | 1 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 10 | 0 | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 14 | 1 | 8 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 7 | 2 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 0 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 6 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 5 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 6 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 6 | 2 | 1 | 2 | 4
Dysgeusia (Nervous system disorders) | 5 | 7 | 0 | 7 | 2
Headache (Nervous system disorders) | 5 | 5 | 1 | 1 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0 | 0 | 4
Anxiety (Psychiatric disorders) | 4 | 3 | 1 | 3 | 1
Confusional state (Psychiatric disorders) | 2 | 1 | 0 | 2 | 2
Insomnia (Psychiatric disorders) | 4 | 9 | 1 | 3 | 4
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 0 | 5 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 1 | 3 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 3
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 3 | 7 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 2 | 8 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 1 | 6 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 0 | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 2 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 2 | 3 | 4
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 3 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 16 | 12 | 2 | 20 | 18
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 19 | 2 | 15 | 14
Erythema (Skin and subcutaneous tissue disorders) | 12 | 10 | 1 | 7 | 3
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 5 | 0 | 4 | 6
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 13 | 3 | 13 | 17
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 28 | 29 | 5 | 25 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 8 | 1 | 8 | 7
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 | 8 | 0 | 5 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 6 | 1 | 9 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 2 | 0
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Hyperaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 9 | 3 | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less